CLINICAL TRIAL: NCT06388304
Title: Pilot Study of Positive Affect Training for Endocrine Therapy Medication Adherence
Brief Title: THRIVE Study: Positive Affect Training for Endocrine Therapy Medication Adherence
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joanna Arch (Other)
Responsible Party: Sponsor-Investigator, Joanna Arch, Principal Investigator, University of Colorado, Boulder
Organization: University of Colorado, Boulder (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-0556
Record Dates: First submitted 2024-04-15; First posted 2024-04-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; DCIS
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Program (Experimental): Online program
  Interventions: Behavioral: THRIVE Online PAT Program

INTERVENTIONS:
Behavioral: THRIVE Online PAT Program — Online program: behavioral intervention based on Positive Affect Training (PAT)

SUMMARY:
The purpose of this study is to pilot and refine an online behavioral intervention based on Positive Affect Training (PAT) that aims to increase positive emotional attitudes and decrease negative emotional attitudes toward endocrine therapy (ET, i.e., anti-hormonal medication) and to increase positive affect and decrease negative affect more generally, among post-treatment breast cancer survivors who are prescribed ET to prevent recurrence of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* hormone receptor-positive breast cancer stages 0-3
* have finished primary treatment (chemotherapy/radiation/surgery)
* are prescribed endocrine therapy (ET) currently or within the last two years
* score above specified cut off (range, 0-10) on any of three questions:

  1. How upset are you by having to take anti-hormonal therapy
  2. How bothered are you by the side effects?
  3. How difficult is it for you to take your anti-hormonal medication every day?
* have internet access to complete online assessments and intervention components or agree to use and return a study wifi-activated iPad.

Exclusion Criteria:

* metastatic disease
* Individuals who are unable to interact with the intervention as needed. This includes those who are extremely visually impaired to the degree that they cannot see the screen and interact as required and individuals who cannot read and/or write in English. This is due to the nature of the intervention itself. If a participant is unable to interact with THRIVE as required, they are unlikely to benefit from the intervention or offer insightful feedback that can be used in refining the program.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Acceptability of THRIVE intervention (AIM) | 1 week post-intervention
  Acceptability of Implementation Measure (Weimer et al., 2017)
Feasibility of THRIVE intervention | 1 week post-intervention
  Feasibility of Intervention Measure (Weimer et al., 2017)
Client Satisfaction Survey | 1 week post-intervention
  Satisfaction and feedback on THRIVE intervention

OTHER OUTCOMES:
Adjuvant endocrine therapy medication adherence (patient-reported) | change from baseline (pre) to 1 week post-intervention (post)
  Wilson et al, 2016, validated 3-item measure of adherence to oral medication
Positive and Negative Affect Scales (PANAS) | change from baseline (pre) to 1 week post-intervention (post)
  Scales that assess positive and negative affect, respectively
Emotional attitudes toward adjuvant endocrine therapy | change from baseline (pre) to 1 week post-intervention (post)
  assessed each positive and negative affective attitudes toward (e.g., emotions associated with) adjuvant endocrine therapy on separate scales, from Rosenberg et al, 2015
Patient Health Questionnaire-8 | change from baseline (pre) to 1 week post-intervention (post)
  Depression questionnaire
Generalized Anxiety Disorder-7 | change from baseline (pre) to 1 week post-intervention (post)
  anxiety symptom questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Arch, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour H, Rosenfield D. Positive affect treatment for depression and anxiety: A randomized clinical trial for a core feature of anhedonia. J Consult Clin Psychol. 2019 May;87(5):457-471. doi: 10.1037/ccp0000396. PMID 30998048
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour HJ. Treatment for Anhedonia: A Neuroscience Driven Approach. Depress Anxiety. 2016 Oct;33(10):927-938. doi: 10.1002/da.22490. PMID 27699943
- [Background] Craske MG, Meuret AE, Echiverri-Cohen A, Rosenfield D, Ritz T. Positive affect treatment targets reward sensitivity: A randomized controlled trial. J Consult Clin Psychol. 2023 Jun;91(6):350-366. doi: 10.1037/ccp0000805. Epub 2023 Mar 9. PMID 36892884
- [Background] Arch JJ, Crespi CM, Levin ME, Genung SR, Nealis M, Mitchell JL, Bright EE, Albright K, Magidson JF, Stanton AL. Randomized Controlled Pilot Trial of a Low-Touch Remotely-Delivered Values Intervention to Promote Adherence to Adjuvant Endocrine Therapy Among Breast Cancer Survivors. Ann Behav Med. 2022 Aug 2;56(8):856-871. doi: 10.1093/abm/kaab118. PMID 35323853